CLINICAL TRIAL: NCT01038583
Title: Aspirin in Reducing Events in the Elderly
Acronym: ASPREE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Bayer (Industry); Monash University (Other); Berman Center for Outcomes and Clinical Research (Other); National Institute on Aging (NIA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSR#09-3029; 3U01AG029824-07S2 (NIH)
Record Dates: First submitted 2009-12-21; First posted 2009-12-24 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Functional Disability; Dementia; Heart Disease; Stroke; Cancer; Bleeding; Depression
Keywords: Aspirin; Prevention; Healthy; Over 70 years old; ASPREE; Aspirin in Reducing Events in the Elderly; Australia; Functional disability; Dementia; Heart Disease/ Stroke; Cancer; Bleeding
MeSH Terms: conditions — Dementia; Heart Diseases; Stroke; Neoplasms; Hemorrhage; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Aspirin: 100 mg enteric-coated aspirin
  Interventions: Drug: 100 mg enteric-coated aspirin
- Placebo: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100 mg enteric-coated aspirin — 100 mg enteric-coated aspirin, taken daily
  Groups: Aspirin
Drug: Placebo — 100 mg enteric-coated placebo
  Groups: Placebo

SUMMARY:
ASPREE-XT is a post-treatment, longitudinal observational follow-up study of ASPREE participants [ASPREE Investigator Group, 2013; www.aspree.org; McNeil et al 2017]. Although the ASPREE trial medication was ceased, the study activity was not stopped and ASPREE participants are continuing with scheduled visits and phone calls. An observational follow-up phase (ASPREE-XT), began in January, 2018. This will enable the monitoring of possible delayed effects of aspirin treatment, primarily on cancer incidence, metastases and mortality. In addition to monitoring the incidence of malignancy within the ASPREE cohort, the opportunity will be taken to observe any other residual effects of aspirin on the endpoints being monitored in the cohort. Continuity of contact with study participants is the key to retention of the cohort for any ongoing or future studies.

DETAILED DESCRIPTION:
ASPREE BACKGROUND:

ASPREE (ASPirin in Reducing Events in the Elderly) is a joint US/Australian research project aiming to determine whether low-dose aspirin increases healthy life-span, defined as survival free of dementia and disability. ASPREE began in 2010 and completed recruitment in 2014. It is a randomized, double-blind, placebo-controlled, primary prevention trial of daily 100 mg of aspirin in a population of healthy older people in the United States (US) and Australia with a period of treatment averaging 4.5 years. ASPREE's primary outcome is length of survival free of dementia and disability and has secondary outcomes encompassing the major health issues related to aging. The trial involving 19,114 persons aged 70 and above (65 years and above for US minorities) is distinctive for its large size, methodological rigor and high participant retention rate in both countries.

ASPREE UNIQUE ASPECTS:

1. It is the first large scale trial to incorporate dementia-free and disability-free survival as a primary outcome. This is now recognized as an appropriate goal of treatment in a primary prevention population of this age group. Within a clinical trial context disability-free survival incorporates an estimate of the overall benefits and risks of aspirin in a single outcome measure.
2. It is one of the first primary prevention trials of aspirin to include cancer incidence, metastases or mortality as a pre-specified endpoint. Recent meta-analyses [Rothwell et al 2010, 2011, 2012] suggests that aspirin has a significant chemopreventive effect becoming evident after a period of 4+ years of aspirin treatment, but questions remain about the magnitude of benefit, and whether it applies to treatment of all cancers and to older people.
3. It will provide information about the impact of aspirin on a range of other conditions (e.g, dementia, CVD, stroke, depression, bleeding) where aspirin has been claimed to have benefit (or risks).

The intervention phase of the trial ended in June 2017 after the NIA determined that it was highly unlikely that aspirin would show a benefit on the overall primary outcome within the planned 5-year time frame. The study is now entering a data cleaning and analysis phase and it is anticipated that the primary results were published in September 2018.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* African American and Hispanic persons age 65 or older
* Any person from another ethnic minority group and Caucasian persons age 70 or older
* Willing and able to provide informed consent, and willing to accept the study requirements

Exclusion Criteria:

* A history of a diagnosed cardiovascular event
* A serious intercurrent illness likely to cause death within the next 5 years, such as terminal cancer or obstructive airways disease
* A current or recurrent condition with a high risk of major bleeding, ex: cerebral aneurysm
* Anemia
* Absolute contraindication or allergy to aspirin
* Current participation in a clinical trial
* Current continuous use of aspirin or other anti-platelet drug or anticoagulant for secondary prevention. People with previous use of aspirin for primary prevention may enter the trial, provided they agree to cease existing use of aspirin and understand that they may be subsequently randomly allocated to low dose aspirin or placebo.
* A systolic blood pressure ≥180 mmHg and / or a diastolic blood pressure ≥105 mmHg
* A history of dementia
* Severe difficulty or an inability to perform any one of the 6 Katz ADLs
* Non-compliance to taking pill

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Men and women recruited from the US and Australia.
  * African American and Hispanic persons age 65 or older in the US
  * Any person from another ethnic minority group and Caucasian persons age 70 or older
  * Willing and able to provide informed consent, and willing to accept the study requirements
Sampling Method: Probability Sample
Enrollment: 19114 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is death from any cause or incident, dementia or persistent physical disability. | every 6 months
  Dementia will be diagnosed based on DSM-IV criteria. Significant physical disability will be defined as a confirmed, and persisting for at least 6 months, self-report of 'a lot of difficulty', or 'inability to perform independently' any one of the 6 Katz basic Activities of Daily Living (ADLs).75

SECONDARY OUTCOMES:
All-cause mortality | every 6 months
Fatal and non fatal cardiovascular events including a) coronary heart disease death, b) non-fatal MI, c) fatal and non-fatal stroke and d) any hospitalization for heart failure | every 6 months
Fatal and non-fatal cancer, excluding non-melanoma skin cancer | every 6 months
Dementia | every 6 months
Mild Cognitive Impairment (MCI; assessed using the Modified Mini-Mental State Examination or 3MS 70 and other cognitive function measures - see below) | every 6 months
Physical disability | every 6 months
Major hemorrhagic events | every 6 months
Depression | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Anne Murray, MD, MSc, Principal Investigator — Berman Center for Outcomes and Clinical Research; John McNeil, MBBS, PHD, Principal Investigator — Monash University
Locations (47):
- United States (33):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Howard University, Washington D.C., District of Columbia
  - University of Florida Department of Aging and Geriatrics, Gainesville, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory/ Atlanta VAMC, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Our Lady of the Lake Cancer Center, Baton Rouge, Louisiana
  - LSU Health Sciences- New Orleans, New Orleans, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - LSU Health Sciences- Shreveport, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Detroit Clinical Research Center, Novi, Michigan
  - HealthPartners Research Institute, Minneapolis, Minnesota
  - Phalen Village Clinic, Saint Paul, Minnesota
  - Central Jersey Medical Center, Elizabeth, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Wake Forest University Baptist Medical Center, Greensboro, North Carolina
  - The Brody School of Medicine at ECU, Greenville, North Carolina
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Health Sciences Research Center, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of TX Medical Branch, Galveston, Texas
  - Regional Academic Health Center, Harlingen, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas
- Australia (14):
  - Clinical Trials Unit, The Canberra Hospital, Garran, Australian Capital Territory
  - Illawarra Health and Medical Research Institute, University of Wollongong, Wollongong, New South Wales
  - Discipline of General Practice, School of Population Health, University of Adelaide, Adelaide, South Australia
  - Greater Green Triangle University, Mount Gambier, South Australia
  - University of Tasmania Rural Clinical School, Burnie, Tasmania
  - The Menzies Institute for Medical Research, University of Tasmania, Hobart, Tasmania
  - University of Tasmania Newnham Campus, Launceston, Tasmania
  - Bendigo Regional Clinical School, Bendigo, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Monash Mildura Regional Clinical School, Mildura, Victoria
  - University of Ballarat, Mount Helen, Victoria
  - Monash Gippsland Regional Clinical School, Traralgon, Victoria
  - The South West Alliance of Rural Health (SWARH), Warrnambool, Victoria
  - Gateway Community Health, Wodonga, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Working with ASPREE - for Data Access requests Monitored secure portal - development underway
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2019
Access Criteria: Will be defined in the Working with ASPREE document

REFERENCES:
- [Background] Barker AL, McNeil JJ, Seeman E, Ward SA, Sanders KM, Khosla S, Cumming RG, Pasco JA, Bohensky MA, Ebeling PR, Woods RL, Lockery JE, Wolfe R, Talevski J; ASPREE Investigator Group. A randomised controlled trial of low-dose aspirin for the prevention of fractures in healthy older people: protocol for the ASPREE-Fracture substudy. Inj Prev. 2016 Aug;22(4):297-301. doi: 10.1136/injuryprev-2015-041655. Epub 2015 May 21. PMID 26002770
- [Background] ASPREE Investigator Group. Study design of ASPirin in Reducing Events in the Elderly (ASPREE): a randomized, controlled trial. Contemp Clin Trials. 2013 Nov;36(2):555-64. doi: 10.1016/j.cct.2013.09.014. Epub 2013 Oct 7. PMID 24113028
- [Derived] McQuilten ZK, Thao LTP, Bick AG, Byars S, Chan AT, Ford L, Leichter A, McNeil JJ, Murray AM, Murphy AJ, Orchard SG, Phung J, Ramshaw HS, Singh J, Tonkin AM, Umar A, Wolfe R, Wood EM, Woods RL, Lacaze P, Curtis DJ. Clonal Hematopoiesis and Cardiovascular Disease and Bleeding Risk and the Effectiveness of Aspirin. JAMA Cardiol. 2025 Dec 1;10(12):1257-1266. doi: 10.1001/jamacardio.2025.3756. PMID 41091476
- [Derived] Thao LTP, Nguyen TL, Singh J, Byars SG, Bick AG, Ford L, Gibbs P, McNeil JJ, Murray AM, Orchard SG, Phung J, Umar A, Wood EM, Woods RL, Lacaze P, Chan AT, Curtis DJ, McQuilten ZK, Wolfe R. Low-Dose Aspirin for Individualized Cancer Prevention in Older Adults: A Secondary Analysis of the ASPREE Randomized Clinical Trial. JAMA Oncol. 2025 Nov 1;11(11):1348-1355. doi: 10.1001/jamaoncol.2025.3593. PMID 40996732
- [Derived] Sheets KM, Webb KL, Woods RL, Orchard SG, Beilin L, Fravel MA, Reid CM, Polkinghorne KR, Wolfe R, Zhou Z, Ryan J, Murray AM, Ernst ME. Long-Term Blood Pressure Variability and Physical Performance in Older Adults. J Clin Hypertens (Greenwich). 2025 Sep;27(9):e70139. doi: 10.1111/jch.70139. PMID 40960215
- [Derived] Sultana F, Islam RM, Davis SR. Associations between declining testosterone concentrations and cognitive performance in community-dwelling older Australian women: a prospective cohort study. Climacteric. 2025 Aug 14:1-7. doi: 10.1080/13697137.2025.2539854. Online ahead of print. PMID 40810327
- [Derived] Brodtmann A, Cheng N, Werden E, Neumann J, Robb C, Fitzgerald SM, Wolfe R, Tonkin AM, Orchard SG, Ryan J, Woods RL, Gao C, McNeil JJ. Cognitive trajectories and incident atrial fibrillation in the ASPREE cohort. medRxiv [Preprint]. 2025 Aug 1:2025.08.01.25332579. doi: 10.1101/2025.08.01.25332579. PMID 40766137
- [Derived] Fravel MA, Ernst ME, Woods RL, Orchard SG, Ganjali S, Wetmore JB, Reid C, Ryan J, Polkinghorne KR, Wolfe R, Nelson MR, Zoungas S, Zhou Z. Performance of the American Heart Association PREVENT Cardiovascular Risk Equations in Older Adults. Circ Cardiovasc Qual Outcomes. 2025 Jun;18(6):e011719. doi: 10.1161/CIRCOUTCOMES.124.011719. Epub 2025 Apr 28. PMID 40289804
- [Derived] Ward SA, Storey E, Naughton MT, Wolfe R, Hamilton GS, Law M, Kawasaki R, Abhayaratna WP, Webb KL, O'Donoghue FJ, Gasevic D, Stocks NP, Trevaks RE, Robman LD, Kolbe S, Fitzgerald SM, Orchard SG, Wong TY, McNeil JJ, Reid CM, Sinclair B, Woods RL. Obstructive sleep apnea and cerebral small vessel disease in community-based older people: an aspirin in reducing events in the elderly imaging substudy. Sleep. 2025 Feb 10;48(2):zsae204. doi: 10.1093/sleep/zsae204. PMID 39301859
- [Derived] Zhou Z, Webb KL, Nelson MR, Woods RL, Ernst ME, Murray AM, Chan AT, Tonkin A, Reid CM, Orchard SG, Kirpach B, Shah RC, Stocks N, Broder JC, Wolfe R. Short- and long-term impact of aspirin cessation in older adults: a target trial emulation. BMC Med. 2024 Jul 29;22(1):306. doi: 10.1186/s12916-024-03507-8. PMID 39075484
- [Derived] Wang Y, Islam RM, Hussain SM, McNeil JJ, Davis SR. Associations Between Blood Concentrations of Sex Hormones and Physical Function in Community-Dwelling Older Women: A Prospective Cohort Study. J Gerontol A Biol Sci Med Sci. 2024 Apr 1;79(4):glad287. doi: 10.1093/gerona/glad287. PMID 38157294
- [Derived] Zhou Z, Tonkin AM, Curtis AJ, Murray A, Zhu C, Reid CM, Williamson JD, Ryan J, McNeil JJ, Beilin LJ, Ernst ME, Stocks N, Lacaze P, Shah RC, Woods RL, Wolfe R, Gall S, Zoungas S, Orchard SG, Nelson MR. Low-Density-Lipoprotein Cholesterol and Mortality Outcomes Among Healthy Older Adults: A Post Hoc Analysis of ASPREE Trial. J Gerontol A Biol Sci Med Sci. 2024 Apr 1;79(4):glad268. doi: 10.1093/gerona/glad268. PMID 38038339
- [Derived] Fravel MA, Ernst ME, Woods RL, Beilin L, Zhou Z, Orchard SG, Chowdhury E, Reid CM, Saifuddin Ekram A, Espinoza SE, Nelson MR, Stocks N, Polkinghorne KR, Wolfe R, Ryan J. Long-term blood pressure variability and frailty risk in older adults. J Hypertens. 2024 Feb 1;42(2):244-251. doi: 10.1097/HJH.0000000000003599. Epub 2023 Nov 20. PMID 38009310
- [Derived] Yu C, Bakshi A, Watts GF, Renton AE, Fulton-Howard B, Goate AM, Natarajan P, Chasman DI, Robman L, Woods RL, Guymer R, Wolfe R, Thao LTP, McNeil JJ, Tonkin AM, Nicholls SJ, Lacaze P. Genome-Wide Association Study of Cardiovascular Resilience Identifies Protective Variation in the CETP Gene. J Am Heart Assoc. 2023 Nov 7;12(21):e031459. doi: 10.1161/JAHA.123.031459. Epub 2023 Nov 6. PMID 37929782
- [Derived] Salih A, Ardissino M, Wagen AZ, Bard A, Szabo L, Ryten M, Petersen SE, Altmann A, Raisi-Estabragh Z. Genome-Wide Association Study of Pericardial Fat Area in 28 161 UK Biobank Participants. J Am Heart Assoc. 2023 Nov 7;12(21):e030661. doi: 10.1161/JAHA.123.030661. Epub 2023 Oct 27. PMID 37889180
- [Derived] Islam RM, Bell RJ, Berk M, Handelsman DJ, McNeil JJ, Wolfe R, Woods RL, Davis SR. Associations between low sex hormone concentrations and depression in older women: An observational study. Maturitas. 2023 Oct;176:107822. doi: 10.1016/j.maturitas.2023.107822. Epub 2023 Aug 4. PMID 37591034
- [Derived] McQuilten ZK, Thao LTP, Pasricha SR, Artz AS, Bailey M, Chan AT, Cohen HJ, Lockery JE, Murray AM, Nelson MR, Schneider HG, Wolfe R, Woods RL, Wood EM, McNeil JJ. Effect of Low-Dose Aspirin Versus Placebo on Incidence of Anemia in the Elderly : A Secondary Analysis of the Aspirin in Reducing Events in the Elderly Trial. Ann Intern Med. 2023 Jul;176(7):913-921. doi: 10.7326/M23-0675. Epub 2023 Jun 20. PMID 37335992
- [Derived] Lockery JE, Collyer TA, Woods RL, Orchard SG, Murray A, Nelson MR, Stocks NP, Wolfe R, Moran C, Ernst ME; ASPREE Investigator Group. Potentially inappropriate medication use is associated with increased risk of incident disability in healthy older adults. J Am Geriatr Soc. 2023 Aug;71(8):2495-2505. doi: 10.1111/jgs.18353. Epub 2023 Apr 11. PMID 37039393
- [Derived] Carr PR, Webb KL, Neumann JT, Thao LTP, Beilin LJ, Ernst ME, Fitzgibbon B, Gasevic D, Nelson MR, Newman AB, Orchard SG, Owen A, Reid CM, Stocks NP, Tonkin AM, Woods RL, McNeil JJ. Associations of body size with all-cause and cause-specific mortality in healthy older adults. Sci Rep. 2023 Mar 7;13(1):3799. doi: 10.1038/s41598-023-29586-w. PMID 36882434
- [Derived] Orchard SG, Lockery JE, Broder JC, Ernst ME, Espinoza S, Gibbs P, Wolfe R, Polekhina G, Zoungas S, Loomans-Kropp HA, Woods RL; ASPREE Investigator Group. Association of metformin, aspirin, and cancer incidence with mortality risk in adults with diabetes. JNCI Cancer Spectr. 2023 Mar 1;7(2):pkad017. doi: 10.1093/jncics/pkad017. PMID 36857596
- [Derived] Sultana F, Davis SR, Murray AM, Woods RL, McNeil JJ, Islam RM. Sex hormones, SHBG and cognitive performance among older Australian women: an observational study. Climacteric. 2023 Apr;26(2):121-128. doi: 10.1080/13697137.2023.2166824. Epub 2023 Jan 30. PMID 36716780
- [Derived] Saifuddin Ekram ARM, Espinoza SE, Ernst ME, Ryan J, Beilin L, Stocks NP, Ward SA, McNeil JJ, Shah RC, Woods RL. The Association between Metabolic Syndrome, Frailty and Disability-Free Survival in Healthy Community-dwelling Older Adults. J Nutr Health Aging. 2023;27(1):1-9. doi: 10.1007/s12603-022-1860-2. PMID 36651481
- [Derived] Ekram ARMS, Ryan J, Espinoza SE, Newman AB, Murray AM, Orchard SG, Fitzgerald SM, McNeil JJ, Ernst ME, Woods RL. The Association between Frailty and Dementia-Free and Physical Disability-Free Survival in Community-Dwelling Older Adults. Gerontology. 2023;69(5):549-560. doi: 10.1159/000528984. Epub 2023 Jan 7. PMID 36617406
- [Derived] Zhou Z, Nelson M, Ernst ME, Reid C, McNeil J, Tonkin A; ASPREE Investigator Group. Does Aspirin Prevent Incident Heart Failure in Healthy Older Adults? Examining the Evidence From the ASPREE Trial. Circ Heart Fail. 2022 Jun;15(6):e009511. doi: 10.1161/CIRCHEARTFAILURE.122.009511. Epub 2022 Apr 5. No abstract available. PMID 35727884
- [Derived] Yan MK, Orchard SG, Adler NR, Wolfe R, McLean C, Rodriguez LM, Woods RL, Gibbs P, Chan AT, Haydon A, Mar VJ. Association between hypertension and cutaneous melanoma, and the effect of aspirin: extended follow-up of a large randomised controlled trial. Cancer Epidemiol. 2022 Aug;79:102173. doi: 10.1016/j.canep.2022.102173. Epub 2022 May 11. PMID 35567859
- [Derived] Polkinghorne KR, Wetmore JB, Thao LTP, Wolfe R, Woods RL, Ernst ME, Nelson MR, Reid CM, Shah RC, McNeil JJ, Murray AM. Effect of Aspirin on CKD Progression in Older Adults: Secondary Analysis From the ASPREE Randomized Clinical Trial. Am J Kidney Dis. 2022 Dec;80(6):810-813. doi: 10.1053/j.ajkd.2022.02.019. Epub 2022 Apr 14. No abstract available. PMID 35430328
- [Derived] Neumann JT, Thao LTP, Murray AM, Callander E, Carr PR, Nelson MR, Wolfe R, Woods RL, Reid CM, Shah RC, Newman AB, Williamson JD, Tonkin AM, McNeil JJ; ASPREE investigators. Prediction of disability-free survival in healthy older people. Geroscience. 2022 Jun;44(3):1641-1655. doi: 10.1007/s11357-022-00547-x. Epub 2022 Apr 14. PMID 35420334
- [Derived] Islam RM, Bell RJ, Handelsman DJ, McNeil JJ, Nelson MR, Reid CM, Tonkin AM, Wolfe RS, Woods RL, Davis SR. Associations between blood sex steroid concentrations and risk of major adverse cardiovascular events in healthy older women in Australia: a prospective cohort substudy of the ASPREE trial. Lancet Healthy Longev. 2022 Feb;3(2):e109-e118. doi: 10.1016/S2666-7568(22)00001-0. Epub 2022 Feb 7. PMID 35252940
- [Derived] Neumann JT, Riaz M, Bakshi A, Polekhina G, Thao LTP, Nelson MR, Woods RL, Abraham G, Inouye M, Reid CM, Tonkin AM, McNeil J, Lacaze P. Prognostic Value of a Polygenic Risk Score for Coronary Heart Disease in Individuals Aged 70 Years and Older. Circ Genom Precis Med. 2022 Feb;15(1):e003429. doi: 10.1161/CIRCGEN.121.003429. Epub 2021 Dec 24. PMID 34949098
- [Derived] Yan MK, Wolfe R, Orchard SG, Ernst ME, Mar VJ. Effect of methotrexate on melanoma risk in older adults: Secondary analysis of a randomised controlled trial. Australas J Dermatol. 2022 Feb;63(1):114-115. doi: 10.1111/ajd.13727. Epub 2021 Sep 28. No abstract available. PMID 34581443
- [Derived] Ernst ME, Fravel MA, Webb KL, Wetmore JB, Wolfe R, Chowdhury E, Reid CM, Woods RL, Beilin L, Margolis KL, Murray AM, Polkinghorne KR. Long-Term Blood Pressure Variability and Kidney Function in Participants of the ASPREE Trial. Am J Hypertens. 2022 Feb 1;35(2):173-181. doi: 10.1093/ajh/hpab143. PMID 34519331
- [Derived] Lacaze P, Riaz M, Sebra R, Hooper AJ, Pang J, Tiller J, Polekhina G, Tonkin A, Reid C, Zoungas S, Murray AM, Nicholls S, Watts G, Schadt E, McNeil JJ. Protective lipid-lowering variants in healthy older individuals without coronary heart disease. Open Heart. 2021 Jul;8(2):e001710. doi: 10.1136/openhrt-2021-001710. PMID 34341098
- [Derived] Ernst ME, Ryan J, Chowdhury EK, Margolis KL, Beilin LJ, Reid CM, Nelson MR, Woods RL, Shah RC, Orchard SG, Wolfe R, Storey E, Tonkin AM, Brodtmann A, McNeil JJ, Murray AM. Long-Term Blood Pressure Variability and Risk of Cognitive Decline and Dementia Among Older Adults. J Am Heart Assoc. 2021 Jul 6;10(13):e019613. doi: 10.1161/JAHA.120.019613. Epub 2021 Jun 26. PMID 34176293
- [Derived] Neumann JT, Riaz M, Bakshi A, Polekhina G, Thao LTP, Nelson MR, Woods RL, Abraham G, Inouye M, Reid CM, Tonkin AM, Williamson JD, Donnan GA, Brodtmann A, Cloud GC, McNeil JJ, Lacaze P. Predictive Performance of a Polygenic Risk Score for Incident Ischemic Stroke in a Healthy Older Population. Stroke. 2021 Aug;52(9):2882-2891. doi: 10.1161/STROKEAHA.120.033670. Epub 2021 May 27. PMID 34039031
- [Derived] Lockery JE, Broder JC, Ryan J, Stewart AC, Woods RL, Chong TT, Cloud GC, Murray A, Rigby JD, Shah R, Storey E, Ward SA, Wolfe R, Reid CM, Collyer TA, Ernst ME; ASPREE Investigator Group, ASPREE Investigator Group listed on www.aspree.org. A Cohort Study of Anticholinergic Medication Burden and Incident Dementia and Stroke in Older Adults. J Gen Intern Med. 2021 Jun;36(6):1629-1637. doi: 10.1007/s11606-020-06550-2. Epub 2021 Mar 22. PMID 33754317
- [Derived] Islam RM, Bell RJ, Handelsman DJ, Robinson PJ, Wolfe R, Davis SR; ASPREE Investigator Group. Longitudinal changes over three years in sex steroid hormone levels in women aged 70 years and over. Clin Endocrinol (Oxf). 2021 Mar;94(3):443-448. doi: 10.1111/cen.14401. Epub 2021 Jan 2. PMID 33351205
- [Derived] Ernst ME, Chowdhury EK, Beilin LJ, Margolis KL, Nelson MR, Wolfe R, Tonkin AM, Ryan J, Woods RL, McNeil JJ, Reid CM; ASPREE Investigator Group. Long-Term Blood Pressure Variability and Risk of Cardiovascular Disease Events Among Community-Dwelling Elderly. Hypertension. 2020 Dec;76(6):1945-1952. doi: 10.1161/HYPERTENSIONAHA.120.16209. Epub 2020 Nov 2. PMID 33131315
- [Derived] Lockery JE, Ernst ME, Broder JC, Orchard SG, Murray A, Nelson MR, Stocks NP, Wolfe R, Reid CM, Liew D, Woods RL; ASPREE Investigator Group. Prescription Medication Use in Older Adults Without Major Cardiovascular Disease Enrolled in the Aspirin in Reducing Events in the Elderly (ASPREE) Clinical Trial. Pharmacotherapy. 2020 Oct;40(10):1042-1053. doi: 10.1002/phar.2461. PMID 33078479
- [Derived] Orchard ER, Ward PGD, Chopra S, Storey E, Egan GF, Jamadar SD. Neuroprotective Effects of Motherhood on Brain Function in Late Life: A Resting-State fMRI Study. Cereb Cortex. 2021 Jan 5;31(2):1270-1283. doi: 10.1093/cercor/bhaa293. PMID 33067999
- [Derived] Mahady SE, Margolis KL, Chan A, Polekhina G, Woods RL, Wolfe R, Nelson MR, Lockery JE, Wood EM, Reid C, Ernst ME, Murray A, Thao L, McNeil JJ. Major GI bleeding in older persons using aspirin: incidence and risk factors in the ASPREE randomised controlled trial. Gut. 2021 Apr;70(4):717-724. doi: 10.1136/gutjnl-2020-321585. Epub 2020 Aug 3. PMID 32747412
- [Derived] Orchard SG, Lockery JE, Gibbs P, Polekhina G, Wolfe R, Zalcberg J, Haydon A, McNeil JJ, Nelson MR, Reid CM, Kirpach B, Murray AM, Woods RL; ASPREE Investigator Group. Cancer history and risk factors in healthy older people enrolling in the ASPREE clinical trial. Contemp Clin Trials. 2020 Sep;96:106095. doi: 10.1016/j.cct.2020.106095. Epub 2020 Jul 31. PMID 32739494
- [Derived] Orchard ER, Ward PGD, Sforazzini F, Storey E, Egan GF, Jamadar SD. Relationship between parenthood and cortical thickness in late adulthood. PLoS One. 2020 Jul 28;15(7):e0236031. doi: 10.1371/journal.pone.0236031. eCollection 2020. PMID 32722686
- [Derived] Ward PGD, Orchard ER, Oldham S, Arnatkeviciute A, Sforazzini F, Fornito A, Storey E, Egan GF, Jamadar SD. Individual differences in haemoglobin concentration influence bold fMRI functional connectivity and its correlation with cognition. Neuroimage. 2020 Nov 1;221:117196. doi: 10.1016/j.neuroimage.2020.117196. Epub 2020 Jul 25. PMID 32721510
- [Derived] Ernst ME, Chowdhury EK, Nelson MR, Reid CM, Margolis KL, Beilin L, Stocks NP, Murray AM, Wolfe R, Lockery JE, Orchard SG, Woods RL, McNeil JJ; ASPREE Investigator Group. Antihypertensive medication use and blood pressure control among treated older adults. J Clin Hypertens (Greenwich). 2020 Aug;22(8):1406-1414. doi: 10.1111/jch.13934. Epub 2020 Jul 15. PMID 32667729
- [Derived] Davis SR, Martinez-Garcia A, Robinson PJ, Handelsman DJ, Desai R, Wolfe R, Bell RJ; ASPREE Investigator Group. Estrone Is a Strong Predictor of Circulating Estradiol in Women Age 70 Years and Older. J Clin Endocrinol Metab. 2020 Sep 1;105(9):e3348-54. doi: 10.1210/clinem/dgaa429. PMID 32614391
- [Derived] Berk M, Woods RL, Nelson MR, Shah RC, Reid CM, Storey E, Fitzgerald S, Lockery JE, Wolfe R, Mohebbi M, Dodd S, Murray AM, Stocks N, Fitzgerald PB, Mazza C, Agustini B, McNeil JJ. Effect of Aspirin vs Placebo on the Prevention of Depression in Older People: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Oct 1;77(10):1012-1020. doi: 10.1001/jamapsychiatry.2020.1214. PMID 32492080
- [Derived] Ryan J, Storey E, Murray AM, Woods RL, Wolfe R, Reid CM, Nelson MR, Chong TTJ, Williamson JD, Ward SA, Lockery JE, Orchard SG, Trevaks R, Kirpach B, Newman AB, Ernst ME, McNeil JJ, Shah RC; ASPREE Investigator Group. Randomized placebo-controlled trial of the effects of aspirin on dementia and cognitive decline. Neurology. 2020 Jul 21;95(3):e320-e331. doi: 10.1212/WNL.0000000000009277. Epub 2020 Mar 25. PMID 32213642
- [Derived] Ryan J, Woods RL, Murray AM, Shah RC, Britt CJ, Reid CM, Wolfe R, Nelson MR, Lockery JE, Orchard SG, Trevaks RE, Chong TJ, McNeil JJ, Storey E; ASPREE Investigator Group. Normative performance of older individuals on the Hopkins Verbal Learning Test-Revised (HVLT-R) according to ethno-racial group, gender, age and education level. Clin Neuropsychol. 2021 Aug;35(6):1174-1190. doi: 10.1080/13854046.2020.1730444. Epub 2020 Feb 26. PMID 32100619
- [Derived] Lockery JE, Rigby J, Collyer TA, Stewart AC, Woods RL, McNeil JJ, Reid CM, Ernst ME; ASPREE Investigator Group. Optimising medication data collection in a large-scale clinical trial. PLoS One. 2019 Dec 27;14(12):e0226868. doi: 10.1371/journal.pone.0226868. eCollection 2019. PMID 31881040
- [Derived] Chowdhury EK, Nelson MR, Ernst ME, Margolis KL, Beilin LJ, Johnston CI, Woods RL, Murray AM, Wolfe R, Storey E, Shah RC, Lockery JE, Tonkin AM, Newman AB, Williamson JD, Abhayaratna WP, Stocks NP, Fitzgerald SM, Orchard SG, Trevaks RE, Donnan GA, Grimm R, McNeil JJ, Reid CM; ASPREE Investigator Group. Factors Associated With Treatment and Control of Hypertension in a Healthy Elderly Population Free of Cardiovascular Disease: A Cross-sectional Study. Am J Hypertens. 2020 Apr 1;33(4):350-361. doi: 10.1093/ajh/hpz192. PMID 31807750
- [Derived] McNeil JJ, Wolfe R, Woods RL, Tonkin AM, Donnan GA, Nelson MR, Reid CM, Lockery JE, Kirpach B, Storey E, Shah RC, Williamson JD, Margolis KL, Ernst ME, Abhayaratna WP, Stocks N, Fitzgerald SM, Orchard SG, Trevaks RE, Beilin LJ, Johnston CI, Ryan J, Radziszewska B, Jelinek M, Malik M, Eaton CB, Brauer D, Cloud G, Wood EM, Mahady SE, Satterfield S, Grimm R, Murray AM; ASPREE Investigator Group. Effect of Aspirin on Cardiovascular Events and Bleeding in the Healthy Elderly. N Engl J Med. 2018 Oct 18;379(16):1509-1518. doi: 10.1056/NEJMoa1805819. Epub 2018 Sep 16. PMID 30221597
- [Derived] McNeil JJ, Woods RL, Nelson MR, Reid CM, Kirpach B, Wolfe R, Storey E, Shah RC, Lockery JE, Tonkin AM, Newman AB, Williamson JD, Margolis KL, Ernst ME, Abhayaratna WP, Stocks N, Fitzgerald SM, Orchard SG, Trevaks RE, Beilin LJ, Donnan GA, Gibbs P, Johnston CI, Ryan J, Radziszewska B, Grimm R, Murray AM; ASPREE Investigator Group. Effect of Aspirin on Disability-free Survival in the Healthy Elderly. N Engl J Med. 2018 Oct 18;379(16):1499-1508. doi: 10.1056/NEJMoa1800722. Epub 2018 Sep 16. PMID 30221596
- [Derived] McNeil JJ, Nelson MR, Woods RL, Lockery JE, Wolfe R, Reid CM, Kirpach B, Shah RC, Ives DG, Storey E, Ryan J, Tonkin AM, Newman AB, Williamson JD, Margolis KL, Ernst ME, Abhayaratna WP, Stocks N, Fitzgerald SM, Orchard SG, Trevaks RE, Beilin LJ, Donnan GA, Gibbs P, Johnston CI, Radziszewska B, Grimm R, Murray AM; ASPREE Investigator Group. Effect of Aspirin on All-Cause Mortality in the Healthy Elderly. N Engl J Med. 2018 Oct 18;379(16):1519-1528. doi: 10.1056/NEJMoa1803955. Epub 2018 Sep 16. PMID 30221595
- [Derived] Margolis KL, Mahady SE, Nelson MR, Ives DG, Satterfield S, Britt C, Ekram S, Lockery J, Schwartz EC, Woods RL, McNeil JJ, Wood EM. Development of a standardized definition for clinically significant bleeding in the ASPirin in Reducing Events in the Elderly (ASPREE) trial. Contemp Clin Trials Commun. 2018 May 22;11:30-36. doi: 10.1016/j.conctc.2018.05.015. eCollection 2018 Sep. PMID 30023457
- [Derived] Ryan J, Woods RL, Britt C, Murray AM, Shah RC, Reid CM, Kirpach B, Wolfe RS, Nelson MR, Lockery JE, Orchard SG, Trevaks RE, McNeil JJ, Storey E; ASPREE Investigator Group. Normative performance of healthy older individuals on the Modified Mini-Mental State (3MS) examination according to ethno-racial group, gender, age, and education level. Clin Neuropsychol. 2019 May;33(4):779-797. doi: 10.1080/13854046.2018.1488996. Epub 2018 Jul 5. PMID 29976121
- [Derived] Wolfe R, Murray AM, Woods RL, Kirpach B, Gilbertson D, Shah RC, Nelson MR, Reid CM, Ernst ME, Lockery J, Donnan GA, Williamson J, McNeil JJ. The aspirin in reducing events in the elderly trial: Statistical analysis plan. Int J Stroke. 2018 Apr;13(3):335-338. doi: 10.1177/1747493017741383. Epub 2017 Nov 7. PMID 29111960
- [Derived] Ward SA, Storey E, Woods RL, Hamilton GS, Kawasaki R, Janke AL, Naughton MT, O'Donoghue F, Wolfe R, Wong TY, Reid CM, Abhayaratna WP, Stocks N, Trevaks R, Fitzgerald S, Hodgson LAB, Robman L, Workman B, McNeil JJ; ASPREE Study Group. The Study of Neurocognitive Outcomes, Radiological and Retinal Effects of Aspirin in Sleep Apnoea- rationale and methodology of the SNORE-ASA study. Contemp Clin Trials. 2018 Jan;64:101-111. doi: 10.1016/j.cct.2017.10.016. Epub 2017 Oct 31. PMID 29097299
- [Derived] Reid CM, Storey E, Wong TY, Woods R, Tonkin A, Wang JJ, Kam A, Janke A, Essex R, Abhayaratna WP, Budge MM; ASPREE Study Group. Aspirin for the prevention of cognitive decline in the elderly: rationale and design of a neuro-vascular imaging study (ENVIS-ion). BMC Neurol. 2012 Feb 8;12:3. doi: 10.1186/1471-2377-12-3. PMID 22315948
- See also: Public ASPREE website — http://www.aspree.org